CLINICAL TRIAL: NCT03971084
Title: Impact of Chewing Gum Containing CPP-ACP on Tooth Mineralisation, Using an in Situ Appliance in Healthy Subjects
Brief Title: Impact of Chewing Gum With CPP-ACP on Tooth Mineralisation in Situ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KBE057
Record Dates: First submitted 2019-05-22; First posted 2019-06-03 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Tooth Demineralization
Keywords: casein phosphopeptide-amorphous calcium phosphate; CPP-ACP; in situ appliance; Transverse Microradiography, TMR; Recaldent; Tooth Remineralization
MeSH Terms: conditions — Tooth Demineralization | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: Monocentric, randomised, double-blind, cross-over controlled study with two arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Same sugar free gum appearance, labelling differ with a letter (A or B)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar free gum without CPP-ACP (Placebo Comparator): Sugar free gum without CPP-ACP, consumed 5 times a day, for 20 min each time, within 5 minutes after 3 main meals plus 2 snacks occasion, during 14 days.
  Interventions: Other: Sugar free gum without CPP-ACP
- Sugar free gum with CPP-ACP (Active Comparator): Sugar free gum with 18.8 mg CPP-ACP per gum, consumed 5 times a day, for 20 min each time, within 5 minutes after 3 main meals plus 2 snacks occasion, during 14 days.
  Interventions: Other: Sugar free gum with CPP-ACP

INTERVENTIONS:
Other: Sugar free gum without CPP-ACP — Sugar free gum without CPP-ACP, consumed 5 times a day, for 20 min each time, within 5 minutes after 3 main meals plus 2 snacks occasion, during 14 days.
  Arms: Sugar free gum without CPP-ACP
Other: Sugar free gum with CPP-ACP — Sugar free gum with 18.8 mg CPP-ACP per gum, consumed 5 times a day, for 20 min each time, within 5 minutes after 3 main meals plus 2 snacks occasion, during 14 days.
  Other Names: Recaldent
  Arms: Sugar free gum with CPP-ACP

SUMMARY:
Monocentric, randomised, double-blind, cross-over controlled study with two arms.

This study aims to analyse the impact on mineralisation of Sugar Free Gum (SFG) containing CPP-ACP in healthy adults.

DETAILED DESCRIPTION:
There is some promising evidence in the literature to support a significant favourable impact of the consumption of Sugar Free Gum (SFG) containing casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) on tooth mineralisation and especially on the promotion of tooth remineralisation, over and above the well-established role of regular SFG, in humans.

This study is a monocentric, randomised, double-blind, cross-over and controlled study. The research hypothesis is that chewing a SFG containing CPP-ACP from Recaldent will better remineralise the enamel in healthy subjects compared with regular SFG, after 2 weeks of gum chewing 5 times a day for 20 minutes within 5 minutes after each meal and snack occasion, with a CPP-ACP dose of 18.8 mg per SFG. This will be studied with an in situ model study, with palatal appliances bearing recessed (1,5mm) human demineralised enamel blocks with caries-like lesions (subsurface lesions), which should be worn 24 h a day by the subjects, including during eating and drinking (but the appliances should be removed for daily oral hygiene procedure and cleaning of the appliance itself). Each appliance will contain two types of the demineralised enamel blocks: half of the blocks will contain shallow subsurface lesions (Carbopol method) and the other half reflecting deeper subsurface lesions (hydroxy-ethyl cellulose method). Both types of lesions have been the subject of oral research interest, as both shallow and deep lesions are involved in caries genesis. Changes in mineralisation of the lesions will be assessed using Transverse Microradiography (TMR).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged between 18 and 55 years old (inclusive)
* Subject has read, signed and received a copy of the Informed Consent prior to initiation of study procedures
* Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits at their appointed time, and to use the product as per instructions
* Subject is in good general health based on medical history and oral soft and hard tissue examination
* Subject with normal salivary flow (unstimulated flow rate ≥0.3ml/min)
* Subject not disliking the taste of the SFG provided
* Subject with stable dietary habits and willing to consume 3 main meals per day with two extra-prandial intakes
* Healthy adults with a BMI value between 20 and 30 kg/m²

Exclusion Criteria:

General criteria

* Subject under legal protection measure
* Subject deprived of liberty by a court or an administrative decision
* Subject currently participating in another study or being in the exclusion period of another study

Biological, therapeutic and medical criteria

* Subject is pregnant, lactating or intend to become pregnant during the course of the clinical study based on oral interview only, as pregnancy may interfere with the outcome of the study
* Subject has a systemic health condition and disorders (such as diabetes HIV positive, AIDS and systemic lupus erythematosis) that could affect the outcome of the study at the discretion of the Investigator
* Any active oral condition, such as caries, periodontal disease, chronic dental neglect or any oral pathology including xerostomia determined by oral evaluation and subject history that in the opinion of the dental examiner could affect the outcome of the study
* Subject has full or partial dentures or any orthodontic appliances (i.e. braces or use of night guards) or tongue or mouth piercing
* Use of other oral care products except the one provided by study team during the wash out period or during the treatment period
* Participation in a research study within the last 30 days
* Subjects treated with antibiotics during the last 30 days or other medications, which in the opinion of the Investigator might influence the study outcome
* Subjects with a history of sensitivity or allergies to ingredients in the study products or allergens present in the production facility (facility which also handles milk, egg, soy, peanut, tree nuts, wheat, fish, crustacean, mollusk, lupine, sesame, seeds, sulphites)Subjects with any concurrent illness, such as a cold, flu, upper respiratory infection, sinusitis or other infectious conditions
* Subjects under a restrictive diet or with a planned weight loss program during the study
* Subjects with severe eating disorders (e.g. anorexia nervosa, binge eating disorder and bulimia)
* Subjects without stable dietary habits or with specific dieting regime, for instance Atkins diet, gluten-free diet and additional specific diets at the discretion of the Investigator
* Subjects who smokes or vapes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Compare the relative mineral weight content measured by Transverse Microradiography (DeltaZd-DeltaZr) on subsurface lesions created by Carbopol method | After 2 weeks intervention period
  Comparison between the 2 groups

SECONDARY OUTCOMES:
Compare the densitometric profile of the demineralised lesion (Delta Zd) measured by Transverse Microradiography on subsurface lesions created by Carbopol method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the densitometric profile of the remineralised lesion (Delta Zr) measured by Transverse Microradiography on subsurface lesions created by Carbopol method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the percent mineral change (%R) measured by Transverse Microradiography on subsurface lesions created by Carbopol method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the lesion depth (LD) measured by Transverse Microradiography on subsurface lesions created by Carbopol method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the change in lesion depth (LDd - LDr) after treatment measured by Transverse Microradiography on subsurface lesions created by Carbopol method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the relative mineral weight content measured by Transverse Microradiography (DeltaZd-DeltaZr) on subsurface lesions created by hydroxy-ethyl cellulose (HEC) method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the densitometric profile of the demineralised lesion (Delta Zd) measured by Transverse Microradiography on subsurface lesions created by hydroxy-ethyl cellulose (HEC) method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the densitometric profile of the remineralised lesion (Delta Zr) measured by Transverse Microradiography on subsurface lesions created by hydroxy-ethyl cellulose (HEC) method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the percent mineral change (%R) measured by Transverse Microradiography on subsurface lesions created by hydroxy-ethyl cellulose (HEC) method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the lesion depth (LD) measured by Transverse Microradiography on subsurface lesions created by hydroxy-ethyl cellulose (HEC) method | After 2 weeks intervention period
  Comparison between the 2 groups
Compare the change in lesion depth (LDd - LDr) after treatment measured by Transverse Microradiography on subsurface lesions created by hydroxy-ethyl cellulose (HEC) method | After 2 weeks intervention period
  Comparison between the 2 groups
Compliance to the number of chewing-gum consumption per day | After 2 weeks intervention period
  Comparison between the 2 groups
Compliance to the length of chewing-gum occasion | After 2 weeks intervention period
  Comparison between the 2 groups
Compliance to the number of meal and snack consumption per day | After 2 weeks intervention period
  Comparison between the 2 groups
Evaluation the compliance to oral appliance wearing (length of appliance wearing per day) | After 2 weeks intervention period
  Comparison between the 2 groups
Evaluation the compliance to oral hygiene compliance: number of oral procedures per day | After 2 weeks intervention period
  Comparison between the 2 groups
Evaluation the compliance to oral hygiene compliance: weight of unused toothpaste | After 2 weeks intervention period
  Comparison between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Higham, Prof., Principal Investigator — The University of Liverpool

IPD SHARING:
Plan to Share IPD: No